CLINICAL TRIAL: NCT01221740
Title: Pain Assessment and Quality of Life in Back Pain Patients: Role of Milnacipran
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decided to discontinue
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Robert N. Jamison, PhD, Robert Jamison, PhD, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-00977/1
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Back Pain
Keywords: To show that patients with greater pain sensitivity; will show greater improvement in their symptoms; (self-reported pain intensity, mood, sleep, and; quality of life) than those with lower pain; sensitivity, based on QST, after taking milnacipran.; To compare outcome differences; (pain intensity, mood, activity interference,; sleep, and side effects) with those patients; who are either taking or not taking opioids for; their pain 10 weeks after being prescribed milnacipran.; To show that patients who are older, male,; with more medical comorbidities, greater disability,; and longer pain duration will report less improvement; (pain, mood, sleep, health-related quality of life); and treatment satisfaction while taking milnacipran; compared with others without such characteristics.; identify patients back or neck pain; greater 6 months; QST; 10 weeks; milnacipran; pain intensity; mood; activity; interference; sleep; side effects; age; gender; medical comorbidities; pain diagnosis; pain duration; disability status
MeSH Terms: conditions — Back Pain; Hypersensitivity; Pain; Neck Pain; Motor Activity; Coitus | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Milnacipran (Experimental): The patients will be titrated to the maintenance dose of 50 mg BID over a 7-day period.
  12.5 mg QD on day 1 12.5 mg BID on days 2 and 3 25 mg BID on days 4, 5, 6, and 7 50 mg BID beginning day 8
  Interventions: Drug: Savella

INTERVENTIONS:
Drug: Savella — The patients will be titrated to the maintenance dose of 50 mg BID over a 7-day period, and will be on the medication for 10 weeks.
  12.5 mg QD on day 1 12.5 mg BID on days 2 and 3 25 mg BID on days 4, 5, 6, and 7 50 mg BID beginning day 8
  Other Names: HCL (Savella), Milnacipran

SUMMARY:
1. To show that patients with greater pain sensitivity will show greater improvement in their symptoms (self-reported pain intensity, mood, sleep, and quality of life) than those with lower pain sensitivity, based on QST, after taking milnacipran.
2. To compare outcome differences (pain intensity, mood, activity interference, sleep, and side effects) with those patients who are either taking or not taking opioids for their pain 10 weeks after being prescribed milnacipran.
3. To show that patients who are older, male, with more medical comorbidities, greater disability, and longer pain duration will report less improvement (pain, mood, sleep, health-related quality of life) and treatment satisfaction while taking milnacipran compared with others without such characteristics.

DETAILED DESCRIPTION:
Chronic pain is a costly syndrome that influences every aspect of a patient's life. Significant interference with sleep, employment, social functioning, and daily activities is common. Chronic pain patients frequently report depression, anxiety, irritability, sexual dysfunction, and decreased energy. Family roles are altered, and worries abound about financial limitations and future consequences of a restricted lifestyle. Epidemiological studies have independently documented that chronic pain is an immense international problem. Chronic pain symptoms afflict one third of the American population (more than 80 million people). Chronic pain accounts for 21% of emergency room visits and 25% of annual missed work days. When direct and indirect costs are considered, chronic pain imposes a greater economic burden than any other disease, with annual estimates up to $100 billion.

Patients will complete a number of questionnaires at baseline and undergo quantitative sensory testing (QST) as well as complete a handheld electronic diary PDA throughout the entire 10 weeks of the study. Patients will be evaluated by a physician and receive a complete history and physical. Radiological studies will be consulted to confirm diagnosis. All subjects who consent to participate in this study will be started on or converted to milnacipran if they are currently taking an SSRI, buproprion, or a TCA. This will be done over a 1 to 2 week period of gradually weaning the antidepressant and escalating milnacipran. All other adjuvant medication will remain constant through the course of the 10-week trial. Efforts will be made to recruit at least 40% of the patients (N= 24) who are not taking opioids for pain.

At the end of the study, all patients will repeat the baseline questionnaires listed above except the demographic questionnaire. They will also be asked to complete the Treatment Helpfulness Questionnaire. We will compare secondary outcome differences (treatment satisfaction and helpfulness) between patients either on or off of opioids.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Primary diagnosis of spinal pain for at least 6 months' duration
* Average pain intensity score of 4 or greater

Exclusion Criteria:

* Current diagnosis of cancer or malignant disease
* Acute bone disease
* History of DSM-IV psychotic disorder
* Pregnancy
* Any illness judged by the PI to interfere with treatment
* Any acute condition requiring surgery
* Currently taking SNRI or MAOI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Decreased Back Pain | Over the course of 10 weeks
  Decreased Back Pain on the Brief Pain Inventory Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital Pain Trials Center, Chestnut Hill, Massachusetts, United States